CLINICAL TRIAL: NCT03606863
Title: A RANDOMIZED, CONTROLLED, CLINICAL TRIAL TO COMPARE PERIPHERAL PARENTERAL NUTRITION (PeriOlimel N4-E) VERSUS CONVENTIONAL FLUID THERAPY IN ENHANCED RECOVERY AFTER SURGERY (ERAS) PROTOCOL IN COLORECTAL CANCER SURGERY.
Brief Title: Peripheral Parenteral Nutrition vs Conventional Fluid in Colorectal Resection in ERAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Antonio Arroyo Sebastian (Other)
Responsible Party: Sponsor-Investigator, Antonio Arroyo Sebastian, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELX-NPP-2016-01
Record Dates: First submitted 2018-07-19; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Colon Cancer; Parenteral Nutrition; Fast-track
MeSH Terms: conditions — Colonic Neoplasms; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perioperative peripheral parenteral nutrition (Experimental): Perioperative peripheral parenteral nutrition during 4 days
  Interventions: Drug: Perioperative peripheral parenteral nutrition
- Standard fluid therapy (No Intervention): Standard fluid therap

INTERVENTIONS:
Drug: Perioperative peripheral parenteral nutrition
  Arms: Perioperative peripheral parenteral nutrition

SUMMARY:
Assess if administration of early nutrition support with Perioperative Peripheral Nutrition (PeriOliclimonel) N4-E) in patients undergoing colon cancer resection in an Enhanced Recovery After Surgery (ERAS) Protocol improve the results of morbi-mortality and hospitalization versus standard intravenous fluid therapy.

DETAILED DESCRIPTION:
The main objective is to determine if perioperative nutritional support with PeriOlimel N4-E, that reaches nutritional requirements of ERAS protocol for colorectal cancer surgery patients, can improve nutritional status so it decreases postoperative complications, hospital length of stay and costs, compared to conventional fluid therapy administration since patients receive oral nutrition at day 3-5.

ELIGIBILITY:
Inclusion Criteria:

* scheduled colorectal cancer surgery
* ASA I-IV

Exclusion Criteria:

* Emergency surgery
* Distant metastasis
* Patient´s refusal to participate
* Allergy or hypersensitivity to egg or soy protein
* Advanced kidney or hepatic impairment
* Severe bleeding disorders
* Congenital abnormalities of amino acid metabolism
* Hyperlipidemia and severe or difficult to control hyperglycemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
morbi-mortality | 30 days
  Early Peripheral Parenteral Nutrition in patients undergoing colon cancer resection in an Enhanced Recovery After Surgery Protocol to improve the results of morbi-mortality and hospitalization versus standard intravenous fluid therapy

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Arroyo, MD, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunidad Valenciana
Locations (1):
- Hospital General Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided